CLINICAL TRIAL: NCT07094178
Title: Efficacy of Corticosteroid Versus Platelet-Rich Plasma Injections in the Treatment of Shoulder Tendinopathy: A Randomized Controlled Trial
Brief Title: Corticosteroid Versus PRP Injections for Shoulder Tendinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Charles Nicolle (Other)
Responsible Party: Principal Investigator, Selma Bouden, assistant doctor, Hopital Charles Nicolle
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRP-CS-2025-CN
Record Dates: First submitted 2025-06-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Tendinopathy of Rotator Cuff
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroid Injection (Experimental): Participants in this arm will receive a single infiltration of corticosteroids into the affected shoulder tendon. Corticosteroids are anti-inflammatory medications commonly used to reduce pain and inflammation in tendinopathies. The injection aims to provide rapid pain relief and improve shoulder function. Patients will be monitored for pain reduction and functional improvement at one week and three months after the injection.
  Interventions: Procedure: Corticosteroid Injection
- Platelet-Rich Plasma (PRP) Injection (Experimental): Participants in this arm will receive a single infiltration of Platelet-Rich Plasma (PRP) into the affected shoulder tendon. PRP is prepared from the patient's own blood and contains growth factors that may promote tissue healing and regeneration. This treatment aims to provide longer-term pain relief and functional improvement. Patients will be evaluated for pain and shoulder function at one week and three months following the injection.
  Interventions: Procedure: platelet-rich plasma injection

INTERVENTIONS:
Procedure: Corticosteroid Injection — This intervention consists of a single injection of corticosteroids administered directly into the affected tendon of the shoulder. Corticosteroids are anti-inflammatory drugs used to rapidly reduce inflammation and pain associated with tendinopathy. The injection is performed under aseptic conditions by a trained physician. The aim is to provide quick pain relief and improve shoulder function, although effects may be temporary.
  Arms: Corticosteroid Injection
Procedure: platelet-rich plasma injection — This intervention involves a single injection of Platelet-Rich Plasma (PRP), which is prepared from the patient's own blood through a process of centrifugation to concentrate platelets. PRP contains growth factors that may promote tissue healing and regeneration. The injection is administered under aseptic conditions into the affected shoulder tendon by a trained physician. The goal is to enhance long-term recovery of tendon function and reduce pain.
  Arms: Platelet-Rich Plasma (PRP) Injection

SUMMARY:
Shoulder tendinopathy is a common condition that causes shoulder pain and limits daily activities. It often results from damage or overuse of the rotator cuff tendons. Treatment typically includes rest, physical therapy, anti-inflammatory medications, and sometimes injections.

This clinical trial aims to compare the effectiveness of two types of injections for treating simple shoulder tendinopathy:

Corticosteroid injections, which reduce inflammation and provide quick pain relief, but may have only short-term effects.

Platelet-Rich Plasma (PRP) injections, a newer treatment made from the patient's own blood, which may promote long-term healing.

The study is being conducted at the Rheumatology Department of Charles Nicolle Hospital in Tunis, Tunisia. A total of 60 adult patients with shoulder tendinopathy will be randomly assigned to receive either a corticosteroid injection or a PRP injection.

Participants will be evaluated before the injection (baseline), after one week, and after three months. The researchers will assess pain levels using a visual analog scale (VAS), and shoulder function using validated questionnaires (DASH and SPADI scores).

The goal is to determine which treatment provides better pain relief and functional improvement over time.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosed with simple tendinopathy of the shoulder confirmed by clinical examination and imaging
* Experiencing shoulder pain for at least 4 weeks
* Able to provide informed consent

Exclusion Criteria:

* Previous shoulder surgery on the affected side
* Presence of rotator cuff tear or severe shoulder pathology
* Systemic inflammatory diseases (e.g., rheumatoid arthritis)
* Recent corticosteroid injection in the affected shoulder (within last 3 months)
* Contraindications to corticosteroids or PRP treatment
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity measured by Visual Analog Scale (VAS) | baseline, 1 week, 3 months
  The Visual Analog Scale (VAS) ranges from 0 to 10, where 0 indicates "no pain" and 10 indicates "worst imaginable pain". Higher scores represent worse pain outcomes.
Change in shoulder function measured by the Disabilities of the Arm, Shoulder and Hand (DASH) score | baseline, 1 week and 3 months
  The DASH score ranges from 0 to 100. Higher scores indicate greater disability (worse function).
Change in shoulder pain and disability measured by the Shoulder Pain and Disability Index (SPADI) | baseline, 1 week, 3 months
  The SPADI score ranges from 0 to 100. Higher scores indicate greater pain and disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Charles Nicolle Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including clinical and demographic data) will be made available to qualified researchers upon reasonable request. Data will be shared after publication of the primary results. Requests can be submitted to the principal investigator, who will review and approve data sharing agreements to ensure participant privacy and compliance with ethical regulations.